CLINICAL TRIAL: NCT03573271
Title: A Prospective, Multi-center, Pivotal Study to Evaluate the Safety and Efficacy of a Micro-Coring Device for the Treatment of Moderate to Severe Facial Wrinkles
Brief Title: Pivotal Study to Evaluate the Effectiveness of a Micro-coring Device Treating Moderate to Severe Facial Wrinkles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cytrellis Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIS 700-00041
Record Dates: First submitted 2018-06-14; First posted 2018-06-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Laxity; Skin
Keywords: facial wrinkles; skin laxity; sagging skin
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Micro-coring of facial/neck skin with MCD (Experimental): Micro coring of facial and neck skin will be conducted in up to 2 treatments and followed 90 days post treatment with MCD
  Interventions: Device: MCD

INTERVENTIONS:
Device: MCD — Micro-coring skin removal with automated coring device

SUMMARY:
Study evaluating the effectiveness of a micro-coring device for the treatment of moderate to severe cheek wrinkles.

DETAILED DESCRIPTION:
Up to 60 subjects who meet the Inclusion/Exclusion criteria will be treated. All subjects will be monitored for a period of 90 days after treatments.

Evaluation results will be based in the following:

* Wrinkle severity score assessed using the Lemperle Wrinkle Scale
* Subject Satisfaction Scale
* PI Global Aesthetic Improvement Scale

ELIGIBILITY:
Inclusion Criteria:

* Males and females 40-70 years of age
* Fitzpatrick Skin Type I to IV as judged by the Investigator.
* Cheek areas are at least a score of 3 using the Lemperle Wrinkle Assessment Scale as judged by the Investigator
* Able to provide written informed consent, understand and willing to comply with all study related procedures and follow-up visits

Exclusion Criteria:

* Lesions suspicious for any malignancy or the presence of actinic keratosis, melasma, vitiligo, cutaneous papules/nodules or active inflammatory lesions in the areas to be treated
* History of keloid formation or hypertrophic scarring
* History of trauma or surgery to the treatment areas in the past 6 months
* Scar present in the areas to be treated
* Silicone injections in the areas to be treated
* Injection of dermal fillers, fat or botulinum toxin, as well as any minimally invasive/invasive medical device for skin treatment, in the study treatment areas, within the past 6 months (i.e., dermabrasion, laser, RF devices)
* Active smokers (0.5 pack/day) or having quit within 3 months prior to treatment
* Active, chronic, or recurrent infection
* History of compromised immune system or currently being treated with immunosuppressive agents
* History of sensitivity to analgesic agents, Aquaphor®, topical or local anesthetics (e.g., lidocaine, benzocaine, procaine) or chlorhexidine, povidone-iodine or epinephrine
* Excessive sun exposure and use of tanning beds or tanning creams within 30 days prior to treatment
* Treatment with aspirin or other blood thinning agents within 14 days prior to treatment
* History or presence of any clinically significant bleeding disorder
* Any issue that, at the discretion of the Investigator, would interfere with assessment of safety or efficacy or compromise the subject's ability to participate in the study
* Treatment with an investigational device or agent within 30 days before treatment or during the study period
* Female and pregnant or plan on becoming pregnant during the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-01-15 (Estimated); Study Completion 2019-03-21 (Estimated)

PRIMARY OUTCOMES:
Assess level of wrinkle improvement using the Lemperle Wrinkle Severity Scale at 90 days post treatment | 90 day post treatment
  Assess level of wrinkle improvement from the baseline to 90 day post treatment an Independent Reviewer(s) using the Lemperle Wrinkle Severity Scale

SECONDARY OUTCOMES:
Assess safety profile by recording of adverse events | 90 days
  Adverse events will be recorded throughout the study

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Laser and Skin Surgery Center of Northern California, Sacramento, California
  - Miami Dermatology and Laser Institute, Miami, Florida
  - Laser and Skin Surgery Center of New York, New York, New York
  - The Practice of Brian S. Biesman, M.D, Nashville, Tennessee
  - Dr A Jay Burns Cosmetic Surgery, Dallas, Texas